CLINICAL TRIAL: NCT00003239
Title: Therapy of Early Chronic Phase Chronic Myelogenous Leukemia (CML) With Alpha Interferon (IFN-A), Low-Dose Cytosine Arabinoside (ARA-C), and Homoharringtonine (HHT)
Brief Title: Chemotherapy and Biological Therapy in Treating Patients With Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM97-229; U01CA070172 (NIH); P30CA016672 (NIH); MDA-DM-97229 (Other: UT MD Anderson Cancer Center); MDA-FDR001791; NCI-T97-0105; CDR0000066114 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; Homoharringtonine; HHT; cephalotaxus alkaloid; cytarabine; Interferon Alpha 2-A; Roferon-A; Ara-C; DepotCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interferon-alpha; Interferon alpha-2; Cytarabine; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy with Cytarabine + Homoharringtonine (Experimental): Interferon alfa and cytarabine daily by subcutaneous injection. Homoharringtonine is administered by continuous infusion on days 1-5.
  Interventions: Biological: Recombinant Interferon Alfa; Drug: Cytarabine; Drug: Omacetaxine Mepesuccinate

INTERVENTIONS:
Biological: Recombinant Interferon Alfa — Daily by subcutaneous injection.
  Other Names: Interferon Alpha 2-A; Roferon-A
Drug: Cytarabine — Daily by subcutaneous injection.
  Other Names: Ara-C; DepotCyt; Cytosine Arabinosine Hydrochloride
Drug: Omacetaxine Mepesuccinate — Homoharringtonine is administered by continuous infusion on days 1-5.
  Other Names: CGX-635-CML-202; HHT; Homoharringtonine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining biological therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy with cytarabine and homoharringtonine and biological therapy with interferon alfa in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effectiveness of low dose cytarabine, homoharringtonine, and interferon alfa in stimulating a complete cytogenic response in patients with Philadelphia chromosome positive early chronic phase chronic myelogenous leukemia. II. Evaluate the duration of the cytogenic response in these patients after this treatment. III. Determine differential success rates and analyze results by prognostic subsets (e.g., risk group, splenomegaly, thrombocytosis, age, etc.) in this patient population.

OUTLINE: Patients receive debulking therapy consisting of hydroxyurea until blood count is at proper level. Patients then receive interferon alfa and cytarabine daily by subcutaneous injection. Homoharringtonine is administered by continuous infusion on days 1-5. Treatment continues for 5-7 years in the absence of unacceptable toxicity or disease progression (accelerated or blastic phase CML). If complete remission is achieved, peripheral blood stem cells are collected. Patients are followed every 3 months for the first year and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically confirmed early chronic phase chronic myelogenous leukemia (CML) Diagnosed within 12 months Philadelphia chromosome positive OR bcr positive No late chronic phase, accelerated phase, or blastic phase CML

PATIENT CHARACTERISTICS: Age: 12 and over Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 2 mg/dL Renal: Creatinine less than 2 mg/dL Cardiovascular: No severe heart disease Other: No psychoses Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Less than 1 month of prior interferon alfa Chemotherapy: Less than 1 month of prior cytarabine Prior hydroxyurea allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 1998-03; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Complete Cytogenic Response | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M. Kantarjian, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org